CLINICAL TRIAL: NCT05894668
Title: A Prospective Assessment of the Perioperative Parameter and Treatment Outcomes of Endoscopic Combined Intrarenal Surgery (ECIRS) in Asia
Brief Title: Perioperative Parameter and Treatment Outcomes of ECIRS in Asia
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2023.172
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ECIRS — Endoscopic Combined Intrarenal Surgery

SUMMARY:
This is an observational, international, multicenter, cohort study, prospectively collecting clinical data registry on consecutive patients with urinary stone undergoing ECIRS.

DETAILED DESCRIPTION:
Patients diagnosed with urinary stones and planned for ECIRS in different centres will be recruited for the study. This registry collects clinical data on patients with ECIRS performed, includes baseline information on demography, symptoms, risk factors, and laboratory variables. Treatment information, perioperative outcomes, and follow-up details (up to 3 months after surgery) will also be collected. In summary, it captures patterns of presentation and treatment parameters, as well as perioperative and short-term outcomes of patients managed by ECIRS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urinary calculi
* Undergoing Endoscopic Combined Intrarenal Surgery (ECIRS)
* Agreed to consent for the study

Exclusion Criteria:

* Patients who have ECIRS for other conditions, such as urothelial cancer etc.
* Patients who intraoperative record was incomplete.
* Patients only have either PCNL or ureteroscopy done (not both)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with urinary stones and planned for ECIRS
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Target Stone status | up to 1 year
  The fragmentation rate of target stone
Treatment related complication | Thirty days after the operation
  he 30-day complications will be graded according to the Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
  - North District Hospital, Sheung Shui

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan SW, Ng CF, Man CW, Chung R, Li SK. A report on a randomly sampled questionnaire survey about renal stone disease in Hong Kong. Hong Kong Med J. 2008 Dec;14(6):427-31. PMID 19060340
- [Background] Taguchi K, Cho SY, Ng AC, Usawachintachit M, Tan YK, Deng YL, Shen CH, Gyawali P, Alenezi H, Basiri A, Bou S, Djojodemedjo T, Sarica K, Shi L, Singam P, Singh SK, Yasui T. The Urological Association of Asia clinical guideline for urinary stone disease. Int J Urol. 2019 Jul;26(7):688-709. doi: 10.1111/iju.13957. Epub 2019 Apr 24. PMID 31016804
- [Background] Scoffone CM, Cracco CM, Cossu M, Grande S, Poggio M, Scarpa RM. Endoscopic combined intrarenal surgery in Galdakao-modified supine Valdivia position: a new standard for percutaneous nephrolithotomy? Eur Urol. 2008 Dec;54(6):1393-403. doi: 10.1016/j.eururo.2008.07.073. Epub 2008 Aug 8. PMID 18715696
- [Background] Cracco CM, Scoffone CM. ECIRS (Endoscopic Combined Intrarenal Surgery) in the Galdakao-modified supine Valdivia position: a new life for percutaneous surgery? World J Urol. 2011 Dec;29(6):821-7. doi: 10.1007/s00345-011-0790-0. Epub 2011 Nov 6. PMID 22057344
- [Background] Hamamoto S, Yasui T, Okada A, Taguchi K, Kawai N, Ando R, Mizuno K, Kubota Y, Kamiya H, Tozawa K, Kohri K. Endoscopic combined intrarenal surgery for large calculi: simultaneous use of flexible ureteroscopy and mini-percutaneous nephrolithotomy overcomes the disadvantageous of percutaneous nephrolithotomy monotherapy. J Endourol. 2014 Jan;28(1):28-33. doi: 10.1089/end.2013.0361. Epub 2013 Oct 24. PMID 23987470